CLINICAL TRIAL: NCT03670355
Title: A Phase 1, Randomized Pharmacokinetic and Safety Study of a 90 Day Intravaginal Ring Containing Tenofovir
Brief Title: Pharmacokinetic and Safety Study of a 90 Day Intravaginal Ring Containing Tenofovir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MTN-038; 38460 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Results first posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tenofovir (TFV) Intravaginal Ring (IVR) (Experimental): The TFV IVR will be inserted during the enrollment visit (Day 0) and used continuously for approximately 91 days.
  Interventions: Drug: Tenofovir (TFV) IVR
- Placebo IVR (Placebo Comparator): The placebo IVR will be inserted during the enrollment visit (Day 0) and used continuously for approximately 91 days.
  Interventions: Drug: Placebo IVR

INTERVENTIONS:
Drug: Tenofovir (TFV) IVR — Contains 1.4 g TFV
  Arms: Tenofovir (TFV) Intravaginal Ring (IVR)
Drug: Placebo IVR — Contains placebo
  Arms: Placebo IVR

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) and safety of a 90-day intravaginal ring (IVR) containing tenofovir (TFV).

DETAILED DESCRIPTION:
This study will evaluate the pharmacokinetics (PK) and safety of a 90-day intravaginal ring (IVR) containing tenofovir (TFV) in healthy, HIV-uninfected individuals assigned female sex at birth.

Participants will be randomly assigned to receive an IVR containing either 1.4 g TFV or placebo. The IVR will be inserted at the enrollment visit (Day 0) and used continuously for approximately 91 days.

Additional study visits will occur at Days 1, 7, 14, 28, 42, 56, 91, and 92. Study visits may include behavioral assessments, physical examinations, blood and urine collection, and pelvic and rectal specimen collection.

ELIGIBILITY:
Inclusion Criteria:

* Assigned female sex at birth

  * Note: Participants who are female at birth, who now identify as male, will not be excluded so long as they are not on female-to-male transition therapy.
* Age 18 through 45 years (inclusive) at Screening, verified per site standard operating procedures (SOPs)
* Able and willing to provide written informed consent to be screened for and enrolled in MTN-038
* Able and willing to provide adequate locator information, as defined in site SOPs
* Able to communicate in spoken and written English
* Available for all visits and able and willing to comply with all study procedural requirements
* Willing to abstain from receptive vaginal or anal sexual activities for 72 hours prior to each clinical visit and for 72 hours after biopsy collection
* Willing to use male condoms for penile-vaginal and penile-rectal sexual intercourse for the duration of study participation
* Per participant report, using an effective method of contraception for at least 30 days (inclusive) prior to Enrollment, and intending to continue use of an effective method for the duration of study participation; effective methods include:

  * hormonal methods (except contraceptive vaginal ring)
  * intrauterine device (IUD)
  * sterilization (of participant or partner, as defined in site SOPs)
  * having sex exclusively with individuals assigned female sex at birth
  * sexually abstinent as defined by abstaining from penile-vaginal intercourse for 90 days prior to Enrollment, and intending to remain abstinent for the duration of study participation
* In general good health as determined by the Investigator of Record (IoR)/designee at Screening and Enrollment
* HIV-uninfected based on testing performed at Screening and Enrollment (per protocol algorithm in the study protocol)
* Per participant report at Screening, regular menstrual cycles with at least 21 days between menses

  * Note: This criterion is not applicable to participants who report using a progestin-only method of contraception at Screening (e.g., Depo-Provera or levonorgestrel-releasing IUD) nor to participants using continuous combination oral contraceptive pills, as the absence of regular menstrual cycles is an expected, normal consequence in this context.
* Per participant report at Screening and Enrollment, states a willingness to refrain from inserting any non-study vaginal and rectal products or objects into the vagina or rectum including, but not limited to spermicides, female condoms, diaphragms, intravaginal rings, vaginal or rectal medications, menstrual cups, cervical caps, douches, lubricants, and sex toys (vibrators, dildos, etc.) for the 24 hours preceding the Enrollment Visit and for the duration of study participation.

  * Note: Use of tampons is permitted except for 24 hours prior to clinic visits in which CVF samples are scheduled to be collected.
* Participants over the age of 21 (inclusive) must have documentation of a satisfactory Pap within the past 3 years prior to Enrollment consistent with Grade 0 according to the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 (Dated November 2007) to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017, or satisfactory evaluation with no treatment required of Grade 1 or higher Pap result
* At Screening and Enrollment, agrees not to participate in other research studies involving drugs, medical devices, vaginal or rectal products, or vaccines after the Screening Visit and for the duration of study participation

Exclusion Criteria:

* Pregnant at Screening or Enrollment or plans to become pregnant during the study period

  * Note: A documented negative pregnancy test performed by study staff is required for inclusion; however, a self-reported pregnancy is adequate for exclusion from the study.
* Diagnosed with symptomatic urinary tract infection (UTI) or reproductive tract infection (RTI) at Screening or Enrollment

  * Otherwise eligible participants diagnosed with UTI/RTI during screening will be offered treatment. If treatment is complete and symptoms have resolved within the 45 day screening window, eligible participants may be enrolled.
  * Note: Asymptomatic BV and candidiasis are not exclusionary.
* Diagnosed with an acute sexually transmitted infection (STI) requiring treatment per current Centers for Disease Control and Prevention (CDC) guidelines (http://www.cdc.gov/std/treatment/) at Screening or Enrollment such as gonorrhea, chlamydia, trichomonas, pelvic inflammatory disease, and/or syphilis

  * Note: Genital warts requiring treatment and frequent recurrence of HSV are considered exclusionary; however, infrequent HSV outbreaks are not. Genital warts requiring treatment are defined as those that cause undue burden or discomfort to the participant, including bulky size, unacceptable appearance, or physical discomfort. See MTN-038 Study-Specific Procedures (SSP) Manual for additional information.
* Has a clinically apparent Grade 2 or higher pelvic exam finding (observed by study staff) at Screening or Enrollment. *

  * Note: Cervical bleeding associated with speculum insertion and/or specimen collection judged to be within the range of normal according to the clinical judgment of the IoR/designee is considered expected non-menstrual bleeding and is not exclusionary.
  * Note: Otherwise eligible participants with exclusionary pelvic exam findings may be enrolled/randomized after the findings have improved to a non-exclusionary severity grading or resolved within 45 days of providing informed consent for screening.
* Participant report and/or clinical evidence of any of the following:

  * Known adverse reaction to any of the study products (ever), including polyurethane
  * Chronic and/or recurrent vaginal candidiasis
  * Non-therapeutic injection drug use in the 12 months prior to Enrollment
  * Last pregnancy outcome less than 90 days prior to Enrollment
  * Gynecologic or genital procedure (e.g., tubal ligation, dilation and curettage, piercing) 45 days or less prior to Enrollment

    * Note: Colposcopy and cervical biopsies for evaluation of an abnormal Pap test as well as IUD insertion/removal are not exclusionary.
  * Currently breastfeeding or planning to breastfeed during the study
  * Participation in any other research study involving drugs, medical devices, vaginal or rectal products, or vaccines, in the 60 days prior to Enrollment
* Use of pre-exposure prophylaxis (PrEP) for HIV prevention and/or post-exposure prophylaxis (PEP) for potential HIV exposure within the 3 months prior to Enrollment, and/or anticipated use and/or unwillingness to abstain from PrEP during trial participation
* Has any of the following laboratory abnormalities at Screening Visit:

  * Grade 1 or higher Aspartate aminotransferase (AST) or alanine transaminase (ALT)*
  * Grade 1 or higher Hemoglobin*
  * Calculated creatinine clearance less than 60 mL/min by the Cockcroft-Gault formula
  * Positive Hepatitis B surface antigen result

    * Note: Otherwise eligible participants with an exclusionary laboratory result may be re-tested during the screening process. If a participant is re-tested and a non-exclusionary result is documented within 45 days of providing informed consent for screening, the participant may be enrolled.
* Has any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate the interpretation of study outcome data, or otherwise interfere with achieving the study objectives including any significant uncontrolled active or chronic medical condition.

(*) Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Corrected Version 2.1, July 2017 and/or Addendum 1 (Female Genital Grading Table for Use in Microbicide Studies [Dated November 2007])

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Liu, MD, MPH, Study Chair — San Francisco Department of Public Health
Locations (3):
- United States (3):
  - Alabama CRS, Birmingham, Alabama
  - Bridge HIV CRS, San Francisco, California
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Liu AY, Gundacker H, Richardson B, Chen BA, Hoesley C, van der Straten A, Brown A, Beamer M, Robinson J, Jacobson CE, Scheckter R, Bunge K, Schwartz J, Thurman A, Piper JM, Marzinke MA; MTN-038 Protocol Team for the Microbicide Trials Network. Phase 1 randomized pharmacokinetic and safety study of a 90-day tenofovir vaginal ring in the United States. J Int AIDS Soc. 2024 Mar;27(3):e26223. doi: 10.1002/jia2.26223. PMID 38444118
- [Derived] Hawley I, Song M, Scheckter R, McClure T, Piper J, Chen BA, Hoesley C, Liu AY, van der Straten A. Users' Preferred Characteristics of Vaginal Rings for HIV Prevention: A Qualitative Analysis of Two Phase I Trials. AIDS Res Hum Retroviruses. 2022 Apr;38(4):313-326. doi: 10.1089/AID.2021.0077. Epub 2022 Feb 11. PMID 34969254

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 49 participants were enrolled and randomized in 3 U.S. medical clinic sites from January 2, 2019 until June 25, 2019.
Pre-assignment Details: 49 participants were enrolled in the study and randomized to study product simultaneously.
Period: Overall Study
Arm/Group | Tenofovir (TFV) Intravaginal Ring (IVR) | Placebo IVR
Started | 33 | 16
Completed | 32 | 14
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Unable to comply with study procedures | 0 | 1
Not completed — Participant refused | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenofovir (TFV) Intravaginal Ring (IVR) | Placebo IVR | Total
Number analyzed (Participants) | 33 | 16 | 49
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29.0 [24 to 35] | 27.5 [23 to 35] | 29.0 [24 to 35]
Age, Customized [Count of Participants; unit: Participants] — Age is measured in years.
  Participants
    Missing | 0 | 0 | 0
    18-19 years | 2 | 0 | 2
    20-24 years | 7 | 5 | 12
    25-29 years | 8 | 5 | 13
    30-34 years | 7 | 2 | 9
    35-39 years | 7 | 2 | 9
    40-45 years | 2 | 2 | 4
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 32 | 14 | 46
  Gender Nonconforming/Gender Variant | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 16 | 49
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 31 | 15 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Black or African American | 8 | 3 | 11
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  White | 18 | 8 | 26
  Other | 1 | 0 | 1
  Mixed | 2 | 4 | 6
  Missing | 0 | 0 | 0
Biological Gender of sex partners [Count of Participants; unit: Participants]
  Both Male and Female | 4 | 3 | 7
  Exclusively Female Partners | 3 | 2 | 5
  Exclusively Male Partners | 19 | 9 | 28
  No Sex Partners | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Measurement of TFV Levels in Plasma
Description: TFV concentrations as assessed by drug detection testing in plasma samples collected at multiple timepoints during the study.
Time Frame: Measured through Day 92
Population: This endpoint includes results from samples collected only from participants randomized to the TFV IVR arm. The samples from participants randomized to placebo will not have any TFV concentrations (outcome measure) in their plasma.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Tenofovir (TFV) Intravaginal Ring (IVR)
Number analyzed (Participants) | 33
pg/mL
  Day 1 postdosing | 636.8 (131.2)
  Day 7 postdosing | 1915.9 (102.3)
  Day 14 postdosing: number analyzed (Participants) | 32
  Day 14 postdosing | 3581.5 (114.7)
  Day 28 postdosing: number analyzed (Participants) | 32
  Day 28 postdosing | 5040.7 (235.0)
  Day 56 postdosing: number analyzed (Participants) | 32
  Day 56 postdosing | 7862.3 (139.6)
  Day 91 postdosing: number analyzed (Participants) | 32
  Day 91 postdosing | 1814.6 (612.2)
  Day 91, 4 hours post-removal: number analyzed (Participants) | 32
  Day 91, 4 hours post-removal | 1081.2 (426.9)
  Day 92, 24 hours post-removal: number analyzed (Participants) | 32
  Day 92, 24 hours post-removal | 236.2 (127.4)

2. Primary Outcome: Measurement of TFV Levels in Cervicovaginal Fluid (CVF)
Description: TFV concentrations as assessed by drug detection testing in CVF samples collected at multiple timepoints during the study.
Time Frame: Measured through Day 92
Population: This endpoint includes results from samples collected only from participants randomized to the TFV IVR arm. The samples from participants randomized to placebo will not have any TFV concentrations (outcome measure) in their CVF.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mg
Arm/Group | Tenofovir (TFV) Intravaginal Ring (IVR)
Number analyzed (Participants) | 33
ng/mg
  Day 0, Hour 1 postdosing | 3 (95.3)
  Day 0, Hour 4 postdosing | 6.2 (92.6)
  Day 1 postdosing | 437.8 (75.1)
  Day 7 postdosing | 1468.2 (129.9)
  Day 14 postdosing: number analyzed (Participants) | 32
  Day 14 postdosing | 2006.4 (57.2)
  Day 28 postdosing: number analyzed (Participants) | 32
  Day 28 postdosing | 2011.8 (288.6)
  Day 56 postdosing: number analyzed (Participants) | 31
  Day 56 postdosing | 2817.1 (70.8)
  Day 91 postdosing: number analyzed (Participants) | 32
  Day 91 postdosing | 270.5 (24859.2)
  Day 91, 4 hours post-removal: number analyzed (Participants) | 32
  Day 91, 4 hours post-removal | 41.3 (406784.3)
  Day 92, 24 hours post-removal: number analyzed (Participants) | 32
  Day 92, 24 hours post-removal | 7.2 (85571.4)

3. Primary Outcome: Measurement of TFV Levels in Rectal Fluid
Description: TFV concentrations as assessed by drug detection testing in rectal fluid samples collected at multiple timepoints during the study.
Time Frame: Measured through Day 92
Population: This endpoint includes results from samples collected only from participants randomized to the TFV IVR arm. The samples from participants randomized to placebo will not have any TFV concentrations (outcome measure) in their rectal fluid.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mg
Arm/Group | Tenofovir (TFV) Intravaginal Ring (IVR)
Number analyzed (Participants) | 33
pg/mg
  Day 1 postdosing | 293.6 (1111.0)
  Day 14 postdosing: number analyzed (Participants) | 32
  Day 14 postdosing | 701.8 (583.2)
  Day 28 postdosing: number analyzed (Participants) | 32
  Day 28 postdosing | 898.3 (1355.9)
  Day 56 postdosing: number analyzed (Participants) | 32
  Day 56 postdosing | 1377.3 (475.9)
  Day 91 postdosing: number analyzed (Participants) | 32
  Day 91 postdosing | 460.3 (1093.3)
  Day 91, 4 hours post-removal: number analyzed (Participants) | 32
  Day 91, 4 hours post-removal | 416.7 (4315.6)

4. Primary Outcome: Measurement of TFV Levels in Cervical Tissue
Description: TFV concentrations as assessed by drug detection testing in cervical tissue samples collected at multiple timepoints during the study.
Time Frame: Measured through Day 92
Population: This endpoint includes results from samples collected only from participants randomized to the TFV IVR arm. The samples from participants randomized to placebo will not have any TFV concentrations (outcome measure) in their cervical tissue. In addition, one participant on the TFV IVR arm declined collection of cervical tissue samples and is not included in the number analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mg
Arm/Group | Tenofovir (TFV) Intravaginal Ring (IVR)
Number analyzed (Participants) | 32
ng/mg
  Day 14 postdosing: number analyzed (Participants) | 15
  Day 14 postdosing | 45.9 (11800.2)
  Day 28 postdosing: number analyzed (Participants) | 17
  Day 28 postdosing | 39.1 (322.8)
  Day 56 postdosing: number analyzed (Participants) | 15
  Day 56 postdosing | 37.1 (177.1)
  Day 91 postdosing: number analyzed (Participants) | 17
  Day 91 postdosing | 6.5 (254895.9)

5. Primary Outcome: Measurement of Tenofovir Diphosphate (TFV-DP) Levels in Cervical Tissue
Description: TFV-DP concentrations as assessed by drug detection testing in cervical tissue samples collected at multiple timepoints during the study.
Time Frame: Measured through Day 92
Population: This endpoint includes results from samples collected only from participants randomized to the TFV IVR arm. The samples from participants randomized to placebo will not have any TFV-DP concentrations (outcome measure) in their cervical tissue. In addition, one participant on the TFV IVR arm refused cervical tissue sample collection.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: fmol/mg
Arm/Group | Tenofovir (TFV) Intravaginal Ring (IVR)
Number analyzed (Participants) | 32
fmol/mg
  Day 14 postdosing: number analyzed (Participants) | 14
  Day 14 postdosing | 2679.5 (82.6)
  Day 28 postdosing: number analyzed (Participants) | 17
  Day 28 postdosing | 3217.8 (85.6)
  Day 56 postdosing: number analyzed (Participants) | 15
  Day 56 postdosing | 1892.6 (178.3)
  Day 91 postdosing: number analyzed (Participants) | 17
  Day 91 postdosing | 456.2 (16735.9)

6. Primary Outcome: Proportion of Participants With Grade 2 or Higher Genitourinary Adverse Event
Description: As defined by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017, and/or Addendum 1 (Female Genital [Dated November 2007] Grading Table for Use in Microbicide Studies)
Time Frame: Measured through Day 92
Population: Includes all participants enrolled and randomized to this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir (TFV) Intravaginal Ring (IVR) | Placebo IVR
Number analyzed (Participants) | 33 | 16
Participants | 4 | 4

7. Primary Outcome: Proportion of Participants With Grade 3 or Higher Adverse Event
Description: As defined by the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017
Time Frame: Measured through Day 92
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir (TFV) Intravaginal Ring (IVR) | Placebo IVR
Number analyzed (Participants) | 33 | 16
Participants | 0 | 0

8. Secondary Outcome: Number of Participants Fully Adherent to the Study IVR
Description: Participants were classified as fully adherent if they kept the study ring inserted at all times during the 91 days of study product use, without any product hold (according to the Product Hold Log eCRF) or ever having the ring out (by self-report in the Ring Adherence eCRF). Ring outages could be ring removals or expulsions (voluntary or involuntary).
Time Frame: Measured through Day 92
Population: The analysis includes all enrolled and randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir (TFV) Intravaginal Ring (IVR) | Placebo IVR
Number analyzed (Participants) | 33 | 16
Participants
  Adherent | 28 | 13
  Non-Adherent | 5 | 3

9. Secondary Outcome: Duration Without IVR in Vagina for Participants Not Fully Adherent
Description: This includes only participants considered non-adherent. Participants were classified as fully adherent if they kept the study ring inserted at all times during the 91 days of study product use, without any product hold (according to the Product Hold Log eCRF) or ever having the ring out (by self-report in the Ring Adherence eCRF).
Time Frame: Measured through Day 92
Population: This analysis includes only participants where were not fully adherent.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tenofovir (TFV) Intravaginal Ring (IVR) | Placebo IVR
Number analyzed (Participants) | 5 | 3
hours | 15.2 (23.1) | 10.0 (14.1)

10. Secondary Outcome: Degree to Which Participants Like or Dislike Using the IVR
Description: This outcome uses question J2 "Overall, how much do you like the ring?" from the final product use end visit (PUEV) behavioral questionnaire. This question and one timepoint were prespecified in the Statistical Analysis Plan (SAP) section 9.2 to represent the participants' overall acceptability of the study product. The question response is on a 10-point Likert scale from 1 to 10 with 1 being extremely dislike to 10 being extremely like. A Likert scale score of 5 is neutral.
Time Frame: Measured on the end of study, Day 92, visit.
Population: This outcome includes all participants who completed the final product use end visit (PUEV) behavioral questionnaire with non-missing response to question J2 "Overall, how much do you like the ring?"
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Tenofovir (TFV) Intravaginal Ring (IVR) | Placebo IVR
Number analyzed (Participants) | 33 | 16
Score on a scale | 8 [7 to 9] | 8 [7 to 10]

ADVERSE EVENTS:
Time Frame: Participants are followed for adverse events during study follow-up which was scheduled up to 3 months (92 days) per participant
Description: As described in section 8.3.1 of the protocol document, study participants will be provided instructions for contacting the study site to report any untoward medical occurrences they may experience. Where feasible and medically appropriate, participants will be encouraged to seek evaluation where a study clinician is based. All participants reporting an untoward medical occurrence will be followed clinically until the occurrence resolves (returns to baseline) or stabilizes.
Groups:
- Tenofovir (TFV) Intravaginal Ring (IVR): The TFV IVR will be inserted during the enrollment visit (Day 0) and used continuously for approximately 91 days.Tenofovir (TFV) IVR: Contains 1.4 g TFV
- Placebo IVR: The placebo IVR will be inserted during the enrollment visit (Day 0) and used continuously for approximately 91 days.Placebo IVR: Contains placebo
Arm/Group | Tenofovir (TFV) Intravaginal Ring (IVR) | Placebo IVR
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/16
Other Adverse Events (participants affected / at risk) | 25/33 | 13/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenofovir (TFV) Intravaginal Ring (IVR) (N=33) | Placebo IVR (N=16)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Suprapubic pain (General disorders) | 1 (1) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 6 (9) | 3 (5)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 4 (5) | 2 (2)
Vulvovaginitis (Infections and infestations) | 2 (3) | 0 (0)
Vulvovaginitis trichomonal (Infections and infestations) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vaginal laceration (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Dyspareunia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Pelvic discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine spasm (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 14 (17) | 8 (9)
Vaginal odour (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Vulval ulceration (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal erythema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT03670355/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-30): https://cdn.clinicaltrials.gov/large-docs/55/NCT03670355/SAP_001.pdf